CLINICAL TRIAL: NCT01080287
Title: The Identification and Characterization of Autonomic Dysfunction in Migraineurs With and Without Auras
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 08-778
Record Dates: First submitted 2010-03-02; First posted 2010-03-04 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Migraine
Keywords: autonomic; orthostatic; syncope; biopsy; prevalence of autonomic dysfunction in migraineurs with orthostatic intolerance; characterize autonomic findings utilizing neurocardiac testing, neurophysiological testing and skin biopsies to analyze autonomic fibers in the dermis
MeSH Terms: conditions — Migraine Disorders; Syncope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Migraineurs with & w/out auras having orthostatic intolerance: Subjects between ages 18 and 65, having ICHD-II classification of migraine with or without aura, having symptoms of orthostatic intolerance
- Migraineurs with or without auras: Subjects between ages 18 and 65 having ICHD-II classification of migraine with or without auras

SUMMARY:
This is a study to compare subject response and symptoms resulting from administration of three clinical assessments.

* The 3 assessments are

1. passive upright tilt table testing,
2. quantitative sudomotor axon reflex testing (QSART)and
3. punch biopsy.

The comparison of results will be from two subject groups:

* Group A, the migraine suffering patient with or without aura
* Group B, the migraine suffering patient with or without aura who has diagnosed orthostatic intolerance (i.e.,feeling dizzy or faint when making a body position change).

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65
* male or female
* migraine diagnosis
* may or may not have orthostatic intolerance
* able to demonstrate study understanding and complete informed consent process

Exclusion Criteria:

* subjects who do not meet inclusion criteria
* subjects unable to complete informed consent process

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Migraineurs with and without auras, half having orthostatic intolerance.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic NI, Center for Headache and Pain, Desk T-33, 9500 Euclid Avenue, Cleveland, Ohio, United States

REFERENCES:
- [Background] Low PA, Opfer-Gehrking TL, Textor SC, Benarroch EE, Shen WK, Schondorf R, Suarez GA, Rummans TA. Postural tachycardia syndrome (POTS). Neurology. 1995 Apr;45(4 Suppl 5):S19-25. PMID 7746369
- [Background] Fouad FM, Tadena-Thome L, Bravo EL, Tarazi RC. Idiopathic hypovolemia. Ann Intern Med. 1986 Mar;104(3):298-303. doi: 10.7326/0003-4819-104-3-298. PMID 3511818
- [Background] McCarthy BG, Hsieh ST, Stocks A, Hauer P, Macko C, Cornblath DR, Griffin JW, McArthur JC. Cutaneous innervation in sensory neuropathies: evaluation by skin biopsy. Neurology. 1995 Oct;45(10):1848-55. doi: 10.1212/wnl.45.10.1848. PMID 7477980
- [Background] Headache Classification Subcommittee of the International Headache Society. The International Classification of Headache Disorders: 2nd edition. Cephalalgia. 2004;24 Suppl 1:9-160. doi: 10.1111/j.1468-2982.2003.00824.x. No abstract available. PMID 14979299